CLINICAL TRIAL: NCT02984540
Title: Effect of a Modified Ketogenic-Mediterranean Diet on Alzheimer's Disease
Acronym: BEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00029992
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2020-07

CONDITIONS: Mild Cognitive Impairment; Insulin Resistance
MeSH Terms: conditions — Cognitive Dysfunction; Insulin Resistance | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOW-CARBOHYDRATE DIET (Experimental): The low-carbohydrate diet will consist of a meal plan of less than 20 grams of carbohydrates per day to be consumed over 6 weeks. Foods that provide high levels of healthy fats (preferably low in saturated fats) will be generously included in the diet plan. Various lean meats, fish, and nutrient rich foods that meet the requirement of less than 20 grams total carbohydrates per day will be included in the meal plans. Carbohydrates will be expected to make up less than 10% of total caloric intake. Participants in the low-carbohydrate diet group will receive a supply of extra virgin olive oil at study visits to incorporate into their individualized meal plans.
  Interventions: Other: Low-Carbohydrate Diet
- LOW-FAT DIET (Experimental): The low-fat diet will consist of a low-fat, higher-carbohydrate meal plan to be consumed over 6 weeks. Participants will be encouraged to limit their amount of fat intake to less than 40 grams per day, while eating plentiful fruits, vegetables, and carbohydrates containing adequate fiber. Various lean meats and other sources of protein will be included in the diet plan. Carbohydrates will be expected to make up 50-60% of total caloric intake.
  Interventions: Other: Low-Fat Diet

INTERVENTIONS:
Other: Low-Carbohydrate Diet — Participants assigned to the Modified Ketogenic-Mediterranean Diet will keep their carbohydrate consumption below 20 grams per day throughout the 6-week intervention.
  Arms: LOW-CARBOHYDRATE DIET
Other: Low-Fat Diet — Participants assigned to the Low-Fat Diet will be encouraged to limit their amount of fat intake to <40 grams/day, while eating plentiful fruits, vegetables, and carbohydrates containing adequate fiber.
  Arms: LOW-FAT DIET

SUMMARY:
The purpose of the BEAM study is to compare the effects of a low-carbohydrate diet and a lowfat diet for adults with mild memory loss and adults with pre-diabetes. The data collected will help determine changes in cognitive function, brain structure and function, and levels of certain proteins and hormones in body fluids.

DETAILED DESCRIPTION:
Participants will be enrolled into 1 of 3 study groups. Group 1 will include healthy volunteers with no apparent memory problems, memory complaints or family history of Alzheimer's disease or dementia. This group will complete cognitive assessments, blood and stool sample collection, neuroimaging, and lumbar puncture at week 0 only. Group 1 will NOT take part in the diet study.

Group 2 will have pre-diabetes, but no apparent memory problems that can be observed during cognitive testing. Group 2 will complete an 18-week diet study, with follow-up assessment 6 weeks after final diet completion. Throughout the study the following will also be completed; cognitive assessments, blood and stool sample collection, neuroimaging, and lumbar puncture.

Group 3 will have mild memory problems that are observed during cognitive testing. Group 3 will complete an 18-week diet study, with follow-up assessment 6 weeks after diet final completion. Throughout the study the following will also be completed; cognitive assessments, blood and stool sample collection, neuroimaging, and lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

1. Male or post-menopausal female;
2. Age 50 to 85 years inclusive;
3. Cognitive diagnosis ranged from cognitively normal for "'Healthy' and 'At-Risk'" to mild/moderate cognitive impairment for "MCI/eAD;"
4. Stable medical condition (generally 3 months prior to screening visit) at the discretion of study physician;
5. Stable on medications (generally 4 weeks prior to screening visit) at the discretion of study physician;
6. Able to complete baseline assessments;
7. HbA1c and fasting glucose within the normal (Healthy or MCI/eAD) or pre-diabetic (At-Risk or MCI/eAD) range depending on group.

Exclusion Criteria:

1. Diagnosis of neurodegenerative illness (except for MCI or early AD in the MCI/eAD group);
2. History of a clinically significant stroke;
3. Current evidence or history in past year of focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse;
4. Sensory impairment (i.e.: visual or auditory) that would preclude the participant from participating in the protocol;
5. Diabetes that requires current use of diabetes medications;
6. Current use of cholesterol/lipid lowering medications;
7. Clinically significant elevations in liver function tests;
8. Active neoplastic disease (stable prostate cancer and non-melanoma skin cancer is permissible);
9. History of epilepsy or seizure within past year;
10. Contraindications for MRI (claustrophobia, craniofacial metal implants, pacemakers);
11. Significant medical illness or organ failure, such as uncontrolled hypertension or cardiovascular disease, chronic obstructive pulmonary disease, liver disease, or kidney disease;
12. Use of the following medications: anticonvulsants, drugs with potential interfering CNS effects (other than cholinesterase inhibitors or memantine), medications with significant anticholinergic activity, anti-parkinsonian medications or regular use of narcotic analgesics;
13. If female, menstruation in the past 12 months or hysterectomy and current hormone replacement therapy medication;
14. Major digestive disorders, absorption issues, or surgeries that may be exacerbated by diet changes;
15. Untreated hypothyroidism or B12 deficiency;
16. Participants currently using resveratrol, CoQ10 (coenzyme Q10), coconut oil/other medium chain triglyceride-containing (ie: Axona) supplements, or curcumin will be excluded unless they are willing to discontinue them 2 weeks prior to the start of baseline visits and remain off for study duration.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Change in spinal fluid levels of biomarkers associated with Alzheimer's disease | Baseline CSF measures will be compared to measures obtained six weeks after the initiation of the ketogenic diet and six weeks after initiation of the American Heart Association Diet

SECONDARY OUTCOMES:
Change in memory composite score | Baseline cognitive measures will be compared to measures obtained six weeks after the initiation of the ketogenic diet and six weeks after initiation of the American Heart Association Diet
Change in insulin sensitivity | Baseline metabolic measures will be compared to measures obtained six weeks after the initiation of the ketogenic diet and six weeks after initiation of the American Heart Association Diet
change in 11C acetoacetate PET uptake | Baseline acetoacetate uptake will be compared to measures obtained six weeks after the initiation of the ketogenic diet and six weeks after initiation of the American Heart Association Diet

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brinkley TE, Leng I, Register TC, Neth BJ, Zetterberg H, Blennow K, Craft S. Changes in Adiposity and Cerebrospinal Fluid Biomarkers Following a Modified Mediterranean Ketogenic Diet in Older Adults at Risk for Alzheimer's Disease. Front Neurosci. 2022 Jun 2;16:906539. doi: 10.3389/fnins.2022.906539. eCollection 2022. PMID 35720727